CLINICAL TRIAL: NCT01521962
Title: A Phase 3 Study to Investigate the Efficacy and Safety of SYR-322 When Used in Combination With Insulin Preparation in Subjects With Type 2 Diabetes in Japan
Brief Title: Study of Combination Therapy With SYR-322
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel
Other Study IDs: SYR-322/CCT-901; U1111-1127-1525 (Registry Identifier: WHO); JapicCTI-121736 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2012-01-26; First posted 2012-01-31 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — alogliptin; Insulin

ARMS (2):
- SYR-322 (Alogliptin) QD (Experimental): SYR-322 25 mg, orally.
  Interventions: Drug: Alogliptin
- Insulin (Placebo Comparator): injection
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets
  Other Names: SYR-322
  Arms: SYR-322 (Alogliptin) QD
Drug: Insulin — Insulin injection
  Arms: Insulin

SUMMARY:
To determine the efficacy and safety of SYR-322 (alogliptin) 25-mg, once daily (QD), in patients with diabetes when used in combination with insulin.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is an outpatient.
2. The subject signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.

Exclusion Criteria:

1. The subject has any serious cardiac disease, serious cerebrovascular disorder, or any serious pancreatic or hematological disease.
2. The subject is considered ineligible for the study for any other reason by the investigator or subinvestigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in glycosylated hemoglobin (HbA1c; Japan Diabetes Society value) | Baseline and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Senior Manager, Study Director — Takeda
Locations (33):
- Japan (33):
  - Aomori, Aomori
  - Hirosaki-shi, Aomori
  - Kashiwa-shi, Chiba
  - Kisarazu-shi, Chiba
  - Kitakyushu-shi, Fukuoka
  - Aki-gun, Hiroshima
  - Fukuyama-shi, Hiroshima
  - Nishinomiya-shi, Hyōgo
  - Koga-shi, Ibaraki
  - Ushiku-shi, Ibaraki
  - Kahoku-gun, Ishikawa-ken
  - Hanamaki-shi, Iwate
  - Morioka, Iwate
  - Kagoshima, Kagoshima-ken
  - Satsuma-sendai-shi, Kagoshima-ken
  - Kumamoto, Kumamoto
  - Minamata-shi, Kumamoto
  - Miyazaki, Miyazaki
  - Nigata-shi, Niigata
  - Hirakata-shi, Osaka
  - Osaka, Osaka
  - Osaka-sayama-shi, Osaka
  - Takatsuki-shi, Osaka
  - Yao-shi, Osaka
  - Kuki-shi, Saitama
  - Ōtsu, Shiga
  - Hamamatsu, Shizuoka
  - Shizuoka, Shizuoka
  - Shimotsuke-shi, Tochigi
  - Shinagawa-ku, Tokyo
  - Toyama, Toyama
  - Sagae-shi, Yamagata
  - Yamagata, Yamagata

REFERENCES:
- [Derived] Kaku K, Mori M, Kanoo T, Katou M, Seino Y. Efficacy and safety of alogliptin added to insulin in Japanese patients with type 2 diabetes: a randomized, double-blind, 12-week, placebo-controlled trial followed by an open-label, long-term extension phase. Expert Opin Pharmacother. 2014 Oct;15(15):2121-30. doi: 10.1517/14656566.2014.956722. Epub 2014 Sep 5. PMID 25190226